CLINICAL TRIAL: NCT06540209
Title: Comparison of Effectiveness of Zinc Supplementation With ORS and Bacillus Clausii Versus Zinc With ORS and Saccharomyces Boulardii in Acute Watery Diarrhea in Paediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWD-CHLAHORE
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Acute Watery Diarrhea
MeSH Terms: interventions — clausin peptide, Bacillus clausii; Probiotics; Zinc; ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacillus clausii + zinc+ ORS group (Experimental): Patients received zinc supplementation with ORS and Bacillus clausii
  Interventions: Drug: Bacillus clausii; Drug: Zinc; Drug: ORS
- Saccharomyces boulardii +zinc+ ORS group (Experimental): Patients were given zinc with ORS and Saccharomyces boulardii
  Interventions: Drug: Saccharomyces boulardii; Drug: Zinc; Drug: ORS

INTERVENTIONS:
Drug: Bacillus clausii — Children will be give Bacillus clausii for 5 days
  Other Names: Probiotics
  Arms: Bacillus clausii + zinc+ ORS group
Drug: Saccharomyces boulardii — Children will be give Saccharomyces boulardii for 5 days
  Other Names: Probiotics
  Arms: Saccharomyces boulardii +zinc+ ORS group
Drug: Zinc — Zinc will be given to all children for 5 days
  Other Names: Standard treatment
Drug: ORS — ORS will be given to all children for 5 days
  Other Names: Standard treatment

SUMMARY:
The current study was carried out to directly compare the effectiveness of zinc supplementation with ORS and Bacillus clausii versus zinc with ORS and Saccharomyces boulardii among the local pediatric population presenting with acute watery diarrhea.

DETAILED DESCRIPTION:
The results and importance of effective treatment for acute watery diarrhea in pediatric patients vary throughout the world. Previously, very limited literature was available comparing the efficacy of Bacillus clausii and Saccharomyces boulardii in acute watery diarrhea, providing mixed results. The current study aims to directly compare the effectiveness of zinc supplementation with ORS and Bacillus clausii versus zinc with ORS and Saccharomyces boulardii.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender
* Aged 3 months to 5 years
* With acute watery diarrhea last less fewer than 14 days
* Presenting with mild to moderate dehydration

Exclusion Criteria:

* Patients with a history of blood or pus in their stools
* History of recent antibiotic or probiotic treatment
* Patients with immunodeficiency conditions, acute systemic illnesses, or chronic diarrhea
* Patients with hypersensitivity to Bacillus clausii or Saccharomyces boulardii

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Stool frequency | 5 days
  Number of stools per day
Stool consistency | 5 days
  Graded on a five-point scale as firm, soft, thick liquid, opaque watery, and watery

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Rizwan, FCPS, Principal Investigator — University of Child Health Sciences, The Children's Hospital Lahore, Pakistan; Muhammad Tufail, MBBS, Principal Investigator — University of Child Health Sciences, The Children's Hospital Lahore, Pakistan; Azher Abbas Shah, Principal Investigator — University of Child Health Sciences, The Children's Hospital Lahore, Pakistan
Locations (1):
- University of Child Health Sciences, The Children's Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable request